CLINICAL TRIAL: NCT01987739
Title: A Single Center, Randomized, Double-blind, Double-dummy, Placebo- and Active-controlled, Six-way Crossover Single-dose Study to Evaluate the Relative Abuse Potential of Almorexant in Recreational Central Nervous System (CNS) Depressant Drug Users
Brief Title: Study to Evaluate the Relative Abuse Potential of Almorexant in Recreational Drug Users
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Midnight Pharma, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple
Other Study IDs: AC-057-116
Record Dates: First submitted 2013-11-13; First posted 2013-11-19 (Estimated); Last update posted 2016-02-12 (Estimated); Status verified 2016-02

CONDITIONS: Abuse Potential Study
Keywords: Almorexant; Zolpidem
MeSH Terms: interventions — almorexant; Zolpidem

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- Arm 1 (Experimental): Subjects were randomized to receive single, oral doses of study medication in the sequence ABFCED, where, Treatment A was: 200 mg almorexant; Treatment B was 400 mg almorexant; Treatment C was 1000 mg almorexant; Treatment D was 20 mg zolpidem; Treatment E was 40 mg zolpidem; and Treatment F was placebo. The duration of each Treatment Visit was 1 day/2 nights. Study drug was administered on Day 1 of each Treatment Visit. Each treatment was separated by a washout period of at least 10 days.
  Interventions: Drug: 200 mg almorexant; Drug: 400 mg almorexant; Drug: 1000 mg almorexant; Drug: 20 mg zolpidem; Drug: 40 mg zolpidem; Drug: placebo
- Arm 2 (Experimental): Subjects were randomized to receive single, oral doses of study medication in the sequence BCADFE, where, Treatment A was: 200 mg almorexant; Treatment B was 400 mg almorexant; Treatment C was 1000 mg almorexant; Treatment D was 20 mg zolpidem; Treatment E was 40 mg zolpidem; and Treatment F was placebo. The duration of each Treatment Visit was 1 day/2 nights. Study drug was administered on Day 1 of each Treatment Visit. Each treatment was separated by a washout period of at least 10 days.
  Interventions: Drug: 200 mg almorexant; Drug: 400 mg almorexant; Drug: 1000 mg almorexant; Drug: 20 mg zolpidem; Drug: 40 mg zolpidem; Drug: placebo
- Arm 3 (Experimental): Subjects were randomized to receive single, oral doses of study medication in the sequence CDBEAF, where, Treatment A was: 200 mg almorexant; Treatment B was 400 mg almorexant; Treatment C was 1000 mg almorexant; Treatment D was 20 mg zolpidem; Treatment E was 40 mg zolpidem; and Treatment F was placebo. The duration of each Treatment Visit was 1 day/2 nights. Study drug was administered on Day 1 of each Treatment Visit. Each treatment was separated by a washout period of at least 10 days.
  Interventions: Drug: 200 mg almorexant; Drug: 400 mg almorexant; Drug: 1000 mg almorexant; Drug: 20 mg zolpidem; Drug: 40 mg zolpidem; Drug: placebo
- Arm 4 (Experimental): Subjects were randomized to receive single, oral doses of study medication in the sequence DECFBA, where, Treatment A was: 200 mg almorexant; Treatment B was 400 mg almorexant; Treatment C was 1000 mg almorexant; Treatment D was 20 mg zolpidem; Treatment E was 40 mg zolpidem; and Treatment F was placebo. The duration of each Treatment Visit was 1 day/2 nights. Study drug was administered on Day 1 of each Treatment Visit. Each treatment was separated by a washout period of at least 10 days.
  Interventions: Drug: 200 mg almorexant; Drug: 400 mg almorexant; Drug: 1000 mg almorexant; Drug: 20 mg zolpidem; Drug: 40 mg zolpidem; Drug: placebo
- Arm 5 (Experimental): Subjects were randomized to receive single, oral doses of study medication in the sequence EFDACB, where, Treatment A was: 200 mg almorexant; Treatment B was 400 mg almorexant; Treatment C was 1000 mg almorexant; Treatment D was 20 mg zolpidem; Treatment E was 40 mg zolpidem; and Treatment F was placebo. The duration of each Treatment Visit was 1 day/2 nights. Study drug was administered on Day 1 of each Treatment Visit. Each treatment was separated by a washout period of at least 10 days.
  Interventions: Drug: 200 mg almorexant; Drug: 400 mg almorexant; Drug: 1000 mg almorexant; Drug: 20 mg zolpidem; Drug: 40 mg zolpidem; Drug: placebo
- Arm 6 (Experimental): Subjects were randomized to receive single, oral doses of study medication in the sequence FAEBDC, where, Treatment A was: 200 mg almorexant; Treatment B was 400 mg almorexant; Treatment C was 1000 mg almorexant; Treatment D was 20 mg zolpidem; Treatment E was 40 mg zolpidem; and Treatment F was placebo. The duration of each Treatment Visit was 1 day/2 nights. Study drug was administered on Day 1 of each Treatment Visit. Each treatment was separated by a washout period of at least 10 days.
  Interventions: Drug: 200 mg almorexant; Drug: 400 mg almorexant; Drug: 1000 mg almorexant; Drug: 20 mg zolpidem; Drug: 40 mg zolpidem; Drug: placebo

INTERVENTIONS:
Drug: 200 mg almorexant
Drug: 400 mg almorexant
Drug: 1000 mg almorexant
Drug: 20 mg zolpidem
Drug: 40 mg zolpidem
Drug: placebo

SUMMARY:
This was a six-way crossover study with six single-dose treatment sessions. The profile of acute effects on abuse potential measures of different almorexant doses was compared to that of placebo and two doses of zolpidem

DETAILED DESCRIPTION:
This was a prospective, randomized, double-blind, double-dummy, balanced, placebo and active-controlled, six-way crossover Phase 1 study with six single-dose treatment sessions. The profile of acute effects on pharmacodynamic abuse potential measures of different almorexant doses was compared with that of placebo and two doses of zolpidem.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subjects 18 to 55 years of age, inclusive.
* Recreational drug use with a history of CNS depressant use, defined as at least 10 lifetime occasions of non-medical use of drugs with depressant/sedative properties (e.g., benzodiazepines, barbiturates, gammahydroxybutyric acid (GHB), zopiclone, zolpidem, cannabis, etc.), and at least one instance of non-medical use in the past year.
* Body mass index (BMI) within the range of 18 to 32 kg/m^2, inclusive, and a minimum weight of 50 kg.
* Female subjects of childbearing potential must have been practicing strict sexual abstinence or using a medically acceptable and reliable form of birth control with a failure rate of < 1% per year from at least 1 month prior to Screening (at least 3 months for oral contraceptives) and for at least 1 month after the last study drug administration. Accepted methods of contraception included implants, injectables, combined oral hormonal contraceptives, some intrauterine devices, sexual abstinence, tubal ligation, or vasectomized partner.
* Female subjects of non-childbearing potential must have been amenorrheic for at least 1 year following natural menopause or had a hysterectomy and/or bilateral oophorectomy (as determined by subject medical history).
* Female subjects must have had a negative pregnancy test at Screening and at each admission.
* Must have passed Qualification Visit eligibility criteria.
* Must have been able to speak, read, and understand English sufficiently to understand the nature of the study, to provide written informed consent, and to allow completion of all study assessments.
* Willing and able to abide by all study requirements and restrictions.
* Give voluntary written informed consent to participate in the study.

Exclusion Criteria:

* Received an investigational drug in a clinical trial within 30 days prior to the Screening Visit.
* Drug or alcohol dependence (except nicotine or caffeine) in the past 2 years as defined by the Diagnostic and Statistical Manual of Mental Disorders (DSM-IV), including subjects who had ever been in a drug rehabilitation program (other than treatment for smoking cessation).
* Unwillingness or inability to abstain from recreational drug use as required for the study.
* Positive urine drug screen at admission to Qualification or any Treatment Visit greater than the established threshold value, except for cannabinoids (THC; due to slow release from adipose tissue). If THC was positive, inclusion was at the discretion of the investigator or designee. Subjects with a positive urine drug screen were rescheduled up to 2-times at the investigator's/designee's discretion.
* Positive breath alcohol test at Screening or at any admission.
* Clinically significant abnormalities on physical examination, medical history, 12-lead electrocardiogram (ECG), vital signs, or laboratory tests, including a history or presence of psychiatric, cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, or oncologic disease or any other condition, which in the opinion of the investigator would have jeopardized the safety of the subject or the validity of the study results.
* Previous history of fainting, collapses, syncope, orthostatic hypotension, or vasovagal reactions.
* Use of non-prescription medication, prescription medication, or natural health products (except vitamin or mineral supplements, acceptable forms of birth control, and hormone replacement) within 7 days prior to first drug administration in the Qualification Visit and throughout the study. Up to 1 g per day of acetaminophen was allowed at the discretion of the investigator. Concomitant medication known to inhibit or induce the cytochrome P3A4 isoenzyme was not allowed. Treatment with drugs metabolized by the cytochrome P2D6 isoenzyme was not allowed.
* History of allergy or hypersensitivity to study drugs, related drugs (e.g., benzodiazepines or gamma-aminobutyric acid related drugs) or excipients (including lactose).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2009-09; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Maximum effect (Emax) over 24 h post-dose for "At the moment" Drug Liking Visual Analogue Scale (VAS) score during each Treatment Visit | 24 hours
  Emax was determined on a Drug Liking VAS which assessed positive and negative drug effects (Griffiths 2003, Milovan 2009, Schoedel 2008). VAS items were displayed on two screen images. Using a mouse, the subject positioned the cursor over the small vertical box ("slider") and clicked on it to move it left or right on a scale of 0-100. To register the response, the subject then pressed the "OK" button that appeared below the horizontal line. A score of '0' represented a 'Strong disliking' and a score of '100' represented a 'Strong liking'.

SECONDARY OUTCOMES:
Minimum Effect (Emin) and Time-weighted mean effect (TWMean) over 24 h post-dose for "At the moment" Drug Liking VAS score during each Treatment Visit | 24 hours
  Emin and TWMean were determined on a Drug Liking VAS which assessed positive and negative drug effects (Griffiths 2003, Milovan 2009, Schoedel 2008). VAS items were displayed on two screen images. Using a mouse, the subject positioned the cursor over the small vertical box ("slider") and clicked on it to move it left or right on a scale of 0-100. To register the response, the subject then pressed the "OK" button that appeared below the horizontal line. A score of '0' represented a 'Strong disliking' and a score of '100' represented a 'Strong liking'.
Overall Drug Liking VAS score (Emax, Emin, and arithmetic mean effect of 8 h and 24 h post-dose assessments during each Treatment Visit) | 24 hours
  Overall drug liking was determined on a Drug Liking VAS which assessed positive and negative drug effects (Griffiths 2003, Milovan 2009, Schoedel 2008). VAS items were displayed on two screen images. Using a mouse, the subject positioned the cursor over the small vertical box ("slider") and clicked on it to move it left or right on a scale of 0-100. To register the response, the subject then pressed the "OK" button that appeared below the horizontal line. A score of '0' represented a 'Strong disliking' and a score of '100' represented a 'Strong liking'.
Good/Bad Drug Effects VAS score (Emax, Emin, and TWMean over 24 h post-dose during each Treatment Visit) | 24 hours
  Good/Bad Drug Effects were determined on a Drug Liking VAS which assessed positive and negative drug effects (Griffiths 2003, Milovan 2009, Schoedel 2008). VAS items were displayed on two screen images. Using a mouse, the subject positioned the cursor over the small vertical box ("slider") and clicked on it to move it left or right on a scale of 0-100. To register the response, the subject then pressed the "OK" button that appeared below the horizontal line. A score of '0' represented 'I can feel bad effects' and a score of '100' represented 'I can feel good effects'.
Take Drug Again VAS score (Emax and arithmetic mean of 8 h and 24 h post-dose assessments during each Treatment Visit) | 24 hours
  Take drug again scores were determined on a Drug Liking VAS which assessed positive and negative drug effects (Griffiths 2003, Milovan 2009, Schoedel 2008). VAS items were displayed on two screen images. Using a mouse, the subject positioned the cursor over the small vertical box ("slider") and clicked on it to move it left or right on a scale of 0-100. To register the response, the subject then pressed the "OK" button that appeared below the horizontal line. A score of '0' represented 'Definitely not' and a score of '100' represented 'Definitely so'.
Subjective Drug Value (SDV) (Emax and arithmetic mean of 8 h and 24 h post-dose assessment during each Treatment Visit) | 24 hours
  The SDV measure involved a series of independent, theoretical forced choices between the drug administered and different monetary values. Subjects were asked to choose between receiving another dose of the same drug to take home or an envelope containing a specified amount of money. However, they did not actually receive either the drug or the money offered in the choices. The monetary value of the drug or the envelope ranged from $0.25 to $50.00.
Feeling High VAS score (Emax and TWMean over 24 h post-dose during each Treatment Visit) | 24 hours
  Feeling high scores were determined on a Drug Liking VAS which assessed positive and negative drug effects (Griffiths 2003, Milovan 2009, Schoedel 2008). VAS items were displayed on two screen images. Using a mouse, the subject positioned the cursor over the small vertical box ("slider") and clicked on it to move it left or right on a scale of 0-100. To register the response, the subject then pressed the "OK" button that appeared below the horizontal line. A score of '0' represented 'Definitely not' and a score of '100' represented 'Definitely so'.
Good Drug Effects VAS score (Emax and TWMean over 24 h post-dose during each Treatment Visit) | 24 hours
  Feeling good drug effect scores were determined on a Drug Liking VAS which assessed positive and negative drug effects (Griffiths 2003, Milovan 2009, Schoedel 2008). VAS items were displayed on two screen images. Using a mouse, the subject positioned the cursor over the small vertical box ("slider") and clicked on it to move it left or right on a scale of 0-100. To register the response, the subject then pressed the "OK" button that appeared below the horizontal line. A score of '0' represented 'Definitely not' and a score of '100' represented 'Definitely so'.
Addiction Research Center Inventory (ARCI) Morphine Benzedrine Group (MBG) scale (Emax and TWMean over 24 h postdose during each Treatment Visit) | 24 hours
  Subjects responded by selecting "False" or "True" with a mouse. One point was given for each response that agreed with the scoring direction on the scale (i.e., true items received a score of 1 if the answer was "True", false items received a score of 1 if the answer was "False"). No points were given when the answer was opposite to the scoring direction. The questions and scoring were part of the 49-item ARCI scale.
Bad Drug Effects VAS score (Emax and TWMean over 24 h post-dose during each Treatment Visit) | 24 hours
  Feeling bad drug effect scores were determined on a Drug Liking VAS which assessed positive and negative drug effects (Griffiths 2003, Milovan 2009, Schoedel 2008). VAS items were displayed on two screen images. Using a mouse, the subject positioned the cursor over the small vertical box ("slider") and clicked on it to move it left or right on a scale of 0-100. To register the response, the subject then pressed the "OK" button that appeared below the horizontal line. A score of '0' represented 'Definitely not' and a score of '100' represented 'Definitely so'.
ARCI Lysergic acid diethylamide (LSD) scale (Emax and TWMean over 24 h post-dose during each Treatment Visit | 24 hours
  Subjects responded by selecting "False" or "True" with a mouse. One point was given for each response that agreed with the scoring direction on the scale (i.e., true items received a score of 1 if the answer was "True", false items received a score of 1 if the answer was "False"). No points were given when the answer was opposite to the scoring direction. The questions and scoring were part of the 49-item ARCI scale.
ARCI Pentobarbital Chlorpromazine Alcohol Group (PCAG) scale (Emax and TWMean over 24 h post-dose during each Treatment Visit) | 24 hours
  Subjects responded by selecting "False" or "True" with a mouse. One point was given for each response that agreed with the scoring direction on the scale (i.e., true items received a score of 1 if the answer was "True", false items received a score of 1 if the answer was "False"). No points were given when the answer was opposite to the scoring direction. The questions and scoring were part of the 49-item ARCI scale.
Alertness/Drowsiness VAS score (Emin [drowsiness] and TWMean over 24 h post-dose during each Treatment Visit) | 24 hours
  Alertness/drowsiness scores were determined on a Drug Liking VAS which assessed positive and negative drug effects (Griffiths 2003, Milovan 2009, Schoedel 2008). VAS items were displayed on two screen images. Using a mouse, the subject positioned the cursor over the small vertical box ("slider") and clicked on it to move it left or right on a scale of 0-100. To register the response, the subject then pressed the "OK" button that appeared below the horizontal line. A score of '0' represented 'Very drowsy' and a score of '100' represented 'Very alert'
Bowdle VAS scores (Emax and TWMean over 24 h post-dose during each Treatment Visit) | 24 hours
  The Bowdle VAS [Bowdle 1998] consists of 13 items for which the subjects were asked to rate their current feelings. Each VAS was scored from 0 to 100, with 0 reflecting "not at all" and 100 reflecting "extremely". Lower individual and overall scores indicated fewer psychedelic effects. The scale was adapted for computer presentation and took approximately 3 minutes to complete.
Any Drug Effects VAS score (Emax and TWMean over 24 h post-dose during each Treatment Visit) | 24 hours
  Feeling any drug effects scores were determined on a Drug Liking VAS which assessed positive and negative drug effects (Griffiths 2003, Milovan 2009, Schoedel 2008). VAS items were displayed on two screen images. Using a mouse, the subject positioned the cursor over the small vertical box ("slider") and clicked on it to move it left or right on a scale of 0-100. To register the response, the subject then pressed the "OK" button that appeared below the horizontal line. A score of '0' represented 'Definitely not' and a score of '100' represented 'Definitely so'.
Drug Familiarity VAS score (Hour 12 during each Treatment Visit) | 12 hours
  Drug familiarity score was determined by asking a general question "How familiar was the effect of the drug you most recently received?" Subjects scored familiarity on a VAS scale from 0-100 where 0 was 'Very unfamiliar' and 100 was 'Very familiar'.
Drug Similarity VAS score (Hour 12 during each Treatment Visit) | 12 hours
  Drug similarity scores were determined by asking 'How similar is the drug you most recently received to [each of a specific drug from a customized list of drugs to which the subject was familiar]?". Subjects scored similarity for each drug on a VAS scale from 0-100 where 0 was 'Not at all similar' and 100 was 'Very similar'.

CONTACTS AND LOCATIONS:
Overall Officials: Edward M Sellers, MD, PhD, Principal Investigator — Kendle Early Stage - Toronto